CLINICAL TRIAL: NCT06081400
Title: A Phase II Multicentric, Randomized Trial Assessing Cryoablation Versus Medical Therapy in Desmoid Tumors Progressing After Watchful Waiting
Brief Title: Cryoablation Versus Medical Therapy in Desmoid Tumors Progressing After Watchful Waiting
Acronym: CRYODESMO-02
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Direction Générale de l'Offre des Soins (DGOS) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 7361
Record Dates: First submitted 2023-08-31; First posted 2023-10-13 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Desmoid Tumor
Keywords: Desmoids; Cryoablation; Drug therapy; Cross-Over Studies
MeSH Terms: conditions — Desmoid Tumors | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryoablation (Experimental): One single cryoablation of the desmoid tumor at Day 0
  Interventions: Procedure: Cryoablation
- Medical therapy (Active Comparator): Chemotherapy: at the investigator's discretion: either
  * methotrexate 30mg/m² + vinblastine 6mg/m² (IV infusion) once/week for 6 months, then every other week from months 7 to 12, or
  * vinorelbine : for adults: 90mg/week (per os: 3x30mg, soft capsules) for 12 months. for adolescents: 60mg/m2/week (capped at 90mg/week) for 12 months
  Interventions: Drug: Chemotherapy drug

INTERVENTIONS:
Procedure: Cryoablation — Percutaneous imaging-guided cryoablation
  Arms: Cryoablation
Drug: Chemotherapy drug — Either :
  methotrexate 30mg/m² + vinblastine 6mg/m² (IV infusion) once/week for 6 months, then every other week from months 7 to 12, or vinorelbine : for adults : 90mg/week (per os: 3x30mg, soft capsules) for 12 months; for adolescents: 60mg/m2/week (capped at 90mg/week) for 12 months
  Arms: Medical therapy

SUMMARY:
"Wait & see" is currently the standard of care of recently diagnosed desmoid tumors (DT). In case of progression or symptomatic disease, medical therapy is nowadays widely used including chemotherapy.

Cryoablation has proven to be beneficial for the treatment of large, progressive and symptomatic DT.

This randomized phase II trial aims to compare cryoablation versus medical therapy in DT patients progressing after the "wait & see" period. Moreover, a cross-over design has been anticipated to allow all patients to undergo cryoablation if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Subject (male or female) with extra-peritoneal desmoid tumor (confirmed by prior biopsy by an experienced pathologist within the RRePS network)
* 13 years of age or older
* Measurable viable tumor (according to the mRECIST criteria using MRI. The baseline MRI imaging is mandatory in the 2 months prior to treatment initiation (D0).
* Progressive disease (according to the mRECIST criteria) after the watchful waiting period or significant increase in symptoms requiring an active therapy, as advised in a multidisciplinary sarcoma tumor board
* Tumor deemed accessible for cryoablation procedure by the operator in a type I center. (In pediatric cases, a careful site tumor analysis will be performed with interventional radiologist to ensure for limited consequence of cryoablation in pediatric patients especially regarding growth plates).
* 100 % of destruction of the tumor achievable in one procedure of cryoablation with 1cm security margin according to assessment by referral center (type 1) for cryoablation
* ECOG performance status 0-2 at inclusion visit
* Biological and hematological parameters (neutrophils ≥ 1,5.109/L ; platelet count ≥ 100.109/L ; no significant hemostatic abnormalities) in the 4 weeks prior to treatment initiation (D0)
* Subject able to understand the objectives and risks of the research and to give dated and signed informed consent. For minors, the consent of the 2 parents must be obtained.
* Subject affiliated to a social health insurance plan
* For a woman of childbearing age: negative blood pregnancy test at screening/inclusion visit
* Subject agreeing to use a contraceptive method

Exclusion criteria:

* Intra-peritoneal or multifocal desmoid tumor
* Concurrent or prior use of any antitumor agent for the current desmoid tumor
* Relapse after surgery for desmoid tumor
* Any contraindication including known hypersensitivity to vinorelbine or other vinca-alkaloids, or other constituents to navelbine, to vinblastine, to methotrexate or any excipients, such as, but not limited to current or recent (within 2 weeks) severe infection, severe renal failure, severe hepatic injury, chronic respiratory failure
* Any contraindication including hypersensitivity to gadoteric acid, meglumine or any drug containing gadolinium
* Concomitant treatment with: yellow fever vaccine, prophylactic treatment with phenytoin, trimethoprim, ciprofloxacin, penicillins, probenecid, acetylsalicylic acid, NSAIDs, PPIs, acitretin, azote protoxide, St John's wort
* Any contra-indication for the procedure as stated by the interventional radiologist in terms of tumor size, proximity to neural/vascular structures or adjacent organs at risk making the procedure at unacceptable risk
* Impaired hemostasis, that may interfere with the conduct of the cryoablation
* Contraindication to any form of sedation
* Others contra-indications to MRI
* Pregnancy or breastfeeding
* Concurrent participation in other experimental studies that could affect endpoints of the present study
* Impossibility to give the subject informed information (subject in an emergency situation, patient with comprehension difficulties ...)
* Psychiatric disorders
* Incompetent subject (subject to a legal protection measure: curatorship, guardianship, future protection mandate, family habilitation)

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Rate of non-progressive disease | 12 months after treatment initiation (Day 0+12months)
  Rates of non-progressive disease (sum of complete response (CR), partial response (PR), and stable disease (SD) according to modified RECIST criteria)

SECONDARY OUTCOMES:
Progression-free survival 1 | from treatment initiation to PD or 24 months whichever comes first
  Progression-free survival 1 (PFS1: from the beginning of cryoablation or medical therapy to first disease progression) in cryoablation and medical therapy group
Rate of patients who cross over to the other arm | 24 months after treatment initiation
Rate of complete response | 12 months after treatment initiation and 12 months after cross-over
  Rate of complete response at 12 months in cryoablation and medical therapy group with and without a cross-over treatment
Secondary Progression-free survival 2 | Through study completion, up to 39 months
  Secondary Progression-free survival 2 (PFS 2: from the cross-over to second disease progression) in cryoablation and medical therapy group
Incidence of Treatment-Emergent Adverse Events as assessed by NCI-CTCAE version 5.0 toxicity scale | Through study completion, up to 39 months
  The occurrence of complications and adverse reactions according to the classification of the NCI-CTCAE version 5.0 toxicity scale
QUALITY OF LIFE assessed by EUROQOL EQ 5D before and after treatment | Screening visit, Month 1, Month 2, Month 3, Month 6, Month 9 and Month 12 after treatment initiation
  EUROQOL EQ 5D will be used; score ranging from 1 (good quality of life) to 5 (poor quality of life)
PAIN assessed by brief pain inventory (BPI) before and after treatment | Screening visit, Day 0/Day 1, Month 1, Month 2, Month 3, Month 6, Month 9 and Month 12 after treatment initiation
  BPI will be used; score ranging from 0 (no pain) to 10 (high pain)
Health economics assessment | Through study completion, up to 39 months
  cost and incremental cost utility ratio

CONTACTS AND LOCATIONS:
Overall Officials: Afshin GANGI, MD, PhD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (13):
- France (13):
  - Service d'oncologie/CHU de Besançon, Besançon
  - Service d'Oncologie Médicale, Service de Radiologie Interventionnelle, Institut BERGONNIE, Bordeaux
  - Service d'Oncologie Médicale, Service de Radiologie Interventionnelle-Centre François BACLESSE, Caen
  - Service d'Oncologie Médicale -Centre Georges François LECLERC, Dijon
  - Service d'Oncologie Médicale, Service de Radiologie Interventionnelle-Centre Léon BERARD, Lyon
  - Service d'Oncologie Médicale, service de Radiologie Interventionnelle,CHU de Marseille, Hopital La Timone, Marseille
  - Service de Radiologie-CHU de Nantes, Nantes
  - Service d'Oncologie Médicale-Centre Antoine LACASSAGNE, Nice
  - Service d'Oncologie Médicale, Saint-Herblain
  - Institut de cancérologie Strasbourg Europe (ICANS), Strasbourg
  - Service d'Imagerie Interventionnelle, Hôpitaux Universitaires de Strasbourg , France, 67091, Strasbourg
  - Service d'Oncologie Médicale-Institut Claudius Régaud et Service de Radiologie Interventionnelle, CHU de Toulouse, Toulouse
  - Service d'Oncologie médicale, Service de Radiologie Interventionnelle- Institut Gustave ROUSSY, Villejuif